CLINICAL TRIAL: NCT04443881
Title: Clinical Trial of the Use of Anakinra in Cytokine Storm Syndrome Secondary to Covid-19. A Phase 2/3, Randomized, Open-label, Parallel Group, 2-arm, Multicenter Study Investigating the Efficacy and Safety of Intravenous Administrations of Anakinra, an Interleukin-1(IL-1) Receptor Antagonist, Added to Standard of Care, Versus Standard of Care, in Reducing Hyper-inflammation and Respiratory Distress in Patients With SARS- CoV-2 Infection
Brief Title: Clinical Trial of the Use of Anakinra in Cytokine Storm Syndrome Secondary to Covid-19 (ANA-COVID-GEAS)
Acronym: ANA-COVID-GEAS
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Fundacion Miguel Servet (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ANA-COVID-GEAS
Record Dates: First submitted 2020-06-18; First posted 2020-06-23 (Actual); Last update posted 2021-06-01 (Actual); Status verified 2021-05

CONDITIONS: COVID-19 Pnemonia
Keywords: Covid-19 disease; pneumonia; Cytokine Storm Sindrome; Anti IL-1; Anakinra
MeSH Terms: conditions — Pneumonia | interventions — Interleukin 1 Receptor Antagonist Protein

STUDY DESIGN:
Intervention Model Description: A phase 2/3, randomized, open label, parallel group, 2-arm, multicenter study investigating the efficacy and safety of intravenous administrations of the study drug,
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Anakinra Arm (Experimental): Standard of care plus Anakinra (100mg) administered as 4-times daily i.v. infusions for a maximun of 15 days
  Interventions: Drug: Anakinra 149 MG/ML Prefilled Syringe [Kineret]
- Control Arm (No Intervention): Standard of care

INTERVENTIONS:
Drug: Anakinra 149 MG/ML Prefilled Syringe [Kineret] — Anakinra (100 mg/ 6 hours) i.v infusión during 15 days
  Arms: Anakinra Arm

SUMMARY:
Phase 2/3 randomized, parallel group, 2-arm study (treatment vs. control), investigating the efficacy and safety of intravenous administration of anakinra, an interleukin 1 receptor antagonist ( IL-1), added to standard treatment, compared to standard treatment alone, to reduce hyperinflammation and respiratory distress in patients with SARS-CoV-2 infection.

DETAILED DESCRIPTION:
This protocol has been prepared by the Systemic Autoimmune Diseases Group (GEAS) steering committee from the Spanish Society of Internal Medicine (SEMI) in response to the current urgent situation that are living in Spain because of the COVID-19 pandemic. The GEAS member are experts in the treatment of autoinflammatory diseases and the use of biologic drugs in general, and anakinra in particular. importantly, in Spain, internal medicine physicians are currently involved in the treatment of patients infected with SARS-CoV-2.

The objective of this study is to investigate new possibilities to reduce the number of patients requiring mechanical ventilation. This is intended to address the most urgent need to preserve the access to intense care unit support to the lower possible number of patients and may potentially reduce mortality.

In December 2019, a respiratory condition caused by what was later identified as a new coronavirus (SARS-CoV-2) was detected in Wuhan Province, China. In these four months, the virus has spread throughout the world's population, in more than 100 countries and affecting thousands of people. The WHO declared in March that we were facing a pandemic because of this virus, in which Europe could now be considered the epicenter. The strict containment measures implemented in China, the mass detection of the virus with subsequent isolation of cases and contacts that has been carried out in countries such as Singapore, Taiwan or South Korea seem to have been useful in limiting the virus´ spread. Consequently, in our country, and given the extension of the infection, a state of alarm has been decreed, at least for four weeks. Despite the containment measures, numerous cases are still being diagnosed every day, with an approximate lethality of 3.7%, especially in those considered at risk such as patients over 60 years of age and with comorbidities (Report nº 17. COVID-19 situation in Spain on 27 March 2020. COVID-19 team. SiViES. CNE. CNM. ISCIII).

When SARS-CoV-2 infects the respiratory tract, it causes the disease called COVID-19. From the point of view of the natural evolution of the disease, this can be a mild respiratory syndrome, which will occur in approximately 80% of cases, or a more serious disease, with the appearance of pulmonary infiltrates and in some patients a respiratory distress with rapidly progressive worsening. This second phase, which is only reached by a subgroup of patients, is usually seen in the interval between day 7 and day 10 of the infection from the onset of symptoms. So far, there is no proven explanation for this great variability in its clinical expression.

The treatment used in our country so far is based on the combination of hydroxychloroquine, azithromycin and antiretrovirals (protease inhibitors, lopinavir), based on previous experiences. Several clinical trials are currently underway in Spain: PanCOVID-19 (Azithromycin + Hydroxychloroquine + lopinavir/ritonavir), GS-US-540-5774 (Remdesivir), EFC16844 (Sarilumab) and WA42380 (Tocilizumab) as well as international projects such as Discovery (NCT04315948), Solidarity and REMAP-CAP which include other treatment alternatives such as interferon-beta-1B or Anakinra.

According to recent data from the Chinese cohorts, a subgroup of patients with COVID-19 shows a very marked increase in inflammatory test data, such as lymphopenia, thrombocytopenia, C-reactive protein (CRP) levels, lactate dehydrogenase (LDH), IL6 (> 40 pg / mL) and D-dimer (> 0.28 μg / L), the latter two being predictive of the development of severe pneumonia (sensitivity 93.3%, specificity 96.4%). Accumulating evidence suggests that a subgroup of patients with severe COVID-19 might have a cytokine storm syndrome (CSS). In this group of patients in which this "inflammatory profile" is detected, the damage observed is not a direct consequence of the viral infection (viral necrotizing pneumonia) but rather a secondary hyperimmune response, mainly related to the monocyte/macrophage activation, which has also been observed in autopsy studies and previously in other infections by other types of coronavirus. This CSS is superimoosable to that observed in patients with secondary hemophagocytic lymphohistiocytosis (sHLH), often triggered by viral infections or macrophage activation syndrome (MAS), secondary to systemic and autoinflammatory autoimmune diseases.

In this group of patients there is a significant release of pro-inflammatory cytokines, including interleukin (IL) -1β and IL-6. Of these, IL-1β has a greater pathogenic relevance, given that it promotes the inflammatory cascade and also induces the synthesis of several inflammatory genes such as IL-6 itself, IL-8, MCP-1, COX-2, IκBα, IL-1α, IL-1β and MKP-1. Numerous case reports and case series have been published supporting the use of IL-1β blockade in the MAS. At this time, there is some experience in the treatment of COVID-19 in the subgroup of patients in the inflammatory phase with Tocilizumab (IL-6 receptor blocker), but no controlled studies have been completed as yet. However, IL-6 is not a key molecule in the cytokine storm that triggers MAS.

Anakinra (IL-1Ra) is a recombinant IL-1 receptor antagonist with a very short half-life of 4-6 hours, requiring a daily subcutaneous injection of a 100 mg dose. It has also been shown to reduce levels of other pro-inflammatory cytokines (including IL-6 and IL-18) and acute phase reactants such as PCR and ferritin. Therefore, it has been used in the control of autoinflammatory syndromes and in patients with MAS. In addition, data have been reported from a phase 3 randomized controlled trial of IL-1 blockade with anakinra in sepsis with characteristics of MAS, which showed a significant improvement in the 28-day survival rate (65.4% anakinra vs. 35.3% placebo), with HR for death 0.28 (0.11-0.71, p = 0.0071), with no increased adverse events.

As shown by the data available in the most recent literature generated from the Chinese experience, and by the most recent data made available by the different Spanish hospitals responsible for the management of these patients, hyper- inflammation, caused by a cytokine storm resulting from an exaggerated response of the immune system to the presence of the virus (CSS-like pneumonia), is considered to represent one of the most important negative prognostic factor in patients infected with SARS-CoV-2. The inclusion criteria for COVID-19 used in this protocol is based on the analysis of routine blood chemistry data obtained from patients with SARS-CoV-2 infection. This criterion has been designed with high sensitivity (>90%) for patients who require ICU admission. This constitute the rationale for testing drugs specifically targeted to reduce the cytokine storm.

This protocol has been prepared for the purpose of addressing the current medical emergency, given the severity of the disease and the extremely high number of individuals affected. The objective of this study is to investigate anakinra to reduce the number of patients requiring mechanical ventilation. This is intended to address the most urgent need to preserve the access to intense care unit support to the lower possible number of patients and may potentially reduce mortality.

The potential applicability of the results of this clinical trial, in an extraordinary health emergency such as COVID-19, is obvious. Positive results could help to define the standard treatment of severe COVID-19 pneumonia and have a dramatic impact on both local and global morbidity and mortality. Negative results would constitute very useful scientific evidence for abandoning unfounded empirical approaches and would help redirect resources and efforts in another more promising direction. The expected length of time needed for recruitment is 3-4 weeks, depending on the epidemiological progression of the pandemic in our centers, so results could be available in early May 2020.

Anakinra is a recombinant form of the human IL-Ra, r-metHuIL-1Ra, which is produced by recombinant DNA technology in an E. coli expression system. Therapeutically, anakinra neutralizes the biological activity of IL-1 (IL-1α and IL-1β) by competitively inhibiting its binding to the IL-1RI.

Kineret (anakinra) was first approved for treatment of RA in the US in 2001 and subsequently in the EU/EEA in 2002. In 2012, an sBLA on anakinra for treatment of NOMID was approved in the US. Kineret is also approved for treatment of CAPS (in EU/EEA, Israel and Australia), Still's disease, including SJIA and AOSD (in EU/EEA) and SJIA (in Australia).

The initial IND for anakinra was granted in 1991. The estimated cumulative exposure to anakinra in completed company sponsored clinical studies up to 1 May 2018 is 6404 subject- years, in 8518 subjects with various indications. Anakinra is administered s.c. at doses of 100 mg/day (RA) or in weight-based doses of up to 8 mg/kg/day (NOMID). In clinical studies in sepsis, doses up to 2 mg/kg/hour i.v. over 72 hours were administered to >500 patients and were well tolerated.

ELIGIBILITY:
* Inclusion Criteria:

  * Age 18-80 years.
  * Severe pneumonia COVID-19 defined as:
  * Nasopharyngeal smear with RCP positive for SARS-CoV-2
  * X-Rays (or other technique) pulmonary infiltrates compatible with pneumonia.
  * 1 or more of the following criteria:
  * Ambient air oxygen saturation <= 94% measured with a pulse oximeter.
  * Pa:FiO2 (partial pressure O2/fraction of inspired O2) <=300.
  * Sa:FiO2 (O2 saturation measured with pulse oximeter/ fraction of inspired O2) <=350.
  * High suspicion of CSS that could resemble MAS-like: represented by IL-6 values > 40 pg/mL and/or ferritin >500 ug/L and/or PCR > 30 mg/L (rationale: ≥ 5 upper normal limit) and/or LDH >300 UI/L. We have chosen these parameters because they are implemented in all the participating hospitals, they are a reflection of the cytokine storm and they have also been significant in terms of predicting mortality in patients with COVID-19 (9).
  * Written informed consent. The protocol will be explained to the patient in front of a nurse who will act as a legal witness by signing the document on behalf of the patient.
* Exclusion Criteria:

  * Need for oro-tracheal intubation and/or invasive mechanical ventilation at the start of the study.
  * AST/ALT with values greater than 5 times normal levels.
  * Neutrophils < 1.500 cell/mmc.
  * Platelets < 50.000 cell/mmc.
  * Sepsis or pneumonia documented by other pathogens than SARS-CoV-2.
  * Existence of any life-threatening comorbidity or any other medical condition that, in the investigator's opinion, makes the patient unsuitable for inclusion.
  * Inability to obtain informed consent.
  * Positivity for HBV, HCV or tuberculin test serology.
  * Pregnancy.
  * Use of other previous or concomitant biological treatments. Patients in concomitant treatment with other biologicals that may interfere will be excluded: tocilizumab, canakinumab, TNFalfa inhibitors, JAKiinibs
  * Severe renal dysfunction (estimated glomerular filtration rate ≤ 30 ml / min / 1.73 m2) or receive continuous renal replacement therapy, hemodialysis or peritoneal dialysis.
  * Uncontrolled hypertension (sitting systolic blood pressure > 180 mmHg or diastolic blood pressure > 110 mmHg).
  * Administration of plasma from convalescent patients who have recovered from SARS-CoV-2 infection.
  * History of hypersensitivity or allergy to any component of the study drug.
  * Enrollment in another concurrent intervention clinical trial, or intake of an investigational medication within three months or 5 half-lives prior to inclusion in this study, if deemed to interfere with the objectives of this study as assessed by the investigator.
  * Predictable inability to cooperate with given instructions or study procedures.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 179 (Actual)
Dates: Start 2020-05-08 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Treatment success, defined as number of patients not requiring mechanical ventilation to assess the effect of anakinra in addition to standard treatment on the need for mechanical ventilation in patients with severe COVID-19 and CSS pneumonia. | Day 15
  Treatment success, defined as number of patients not requiring mechanical ventilation by Day 15.
Number of patients not requiring mechanical ventilation to assess the effect of anakinra in addition to standard treatment on the need for mechanical ventilation in patients with severe COVID-19 and CSS pneumonia. | Day 28
  Number of patients not requiring mechanical ventilation
Time to mechanical ventilation to assess the effect of anakinra in addition to standard treatment on the need for mechanical ventilation in patients with severe COVID-19 and CSS pneumonia. | Up to 28 days
  Time to mechanical ventilation
Time to oxygen saturation normalization to assess the effect of anakinra in addition to standard treatment on the need for mechanical ventilation in patients with severe COVID-19 and CSS pneumonia. | Up to 28 days
  Time to oxygen saturation normalization
Stay in ICU and hospitalization to assess the effect of anakinra in addition to standard treatment on the need for mechanical ventilation in patients with severe COVID-19 and CSS pneumonia. | Up to 28 days
  Stay in ICU and hospitalization

SECONDARY OUTCOMES:
Total mortality rate to assess the effect of anakinra in addition to standard treatment on mortality in patients with severe COVID-19 and CSS pneumonia. | day 28
  Total mortality rate
Mortality 48 hours, 7 days, in ICU and hospital to assess the effect of anakinra in addition to standard treatment on mortality in patients with severe COVID-19 and CSS pneumonia. | 48 hours, 7 days
  Mortality 48 hours, 7 days, in ICU and hospital
Viral clearance / viral shedding to assess the effect of anakinra in addition to standard treatment on mortality in patients with severe COVID-19 and CSS pneumonia. | Up to 28 days
  Viral clearance / viral shedding
To assess the effect of anakinra in addition to standard treatment on mortality in patients with severe COVID-19 and CSS pneumonia. | At day 28
  Frequency and severity of AEs: Treatment-emergent severe fatal and life-threatening serious adverse events (SAEs), Adverse events leading to premature discontinuation of study treatment, Anaphylactic/anaphylactoid reactions, Anakinra treatment group: Severe neutropenia, Treatment-emergent laboratory abnormalities.

OTHER OUTCOMES:
Change in IL-6 to assess the effect of anakinra on IL-6, ferritin, and selected biomarkers relevant for hyperinflammation, MAS and cytokine storm change from baseline. | During 28 days
  Change (improvement) in IL-6
Change in ferritin to assess the effect of anakinra | During 28 days
  Change (improvement) in ferritin
Change in D-dimer to assess the effect of anakinra | During 28 days
  Change (improvement) in D-dimer
Change in TGs to assess the effect of anakinra | During 28 days
  Change (improvement) in TGs
Change in lymphopenia to assess the effect of anakinra | During 28 days
  Change (improvement) in lymphopenia
Change in CRP to assess the effect of anakinra | During 28 days
  Change (improvement) in CRP
Change in ESR to assess the effect of anakinra | During 28 days
  Change (improvement) in ESR
Change in LDH to assess the effect of anakinra | During 28 days
  Change (improvement) in LDH
Time to defervescence to assess the effect of anakinra | During 28 days
  Time to defervescence (fever end)

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Fanlo Mateo, PhD, Principal Investigator — Complejo Hospitalario de Navarra
Locations (12):
- Spain (12):
  - Hospital Universitario Miguel Servet, Zaragoza, Aragon
  - Hospital Clinic, Barcelona, Catalonia
  - Hospital Universitario Vall d´Hebron, Barcelona, Catalonia
  - Complexo Hospitalario Universitario de Santiago, Santiago de Compostela, Galicia
  - Hospital Universitario Son Espases, Palma de Mallorca, Mallorca
  - Complejo Hospitalario de Navarra, Pamplona, Navarre
  - Hospital Universitario de Cabueñes, Gijón, Principality of Asturias
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Universitario y Politecnico La Fe, Valencia
  - Complejo Hospitalario Universitario de Vigo, Vigo
  - Hospital Clínico Universitario Lozano Blesa, Zaragoza

IPD SHARING:
Plan to Share IPD: No
All collected IPD will be available for exploitation in future research projects. This statement also includes the availability of the study protocol, the statistical analysis plan, the informed consent form, the clinical study report and the analytic code.

REFERENCES:
- [Derived] Fanlo P, Gracia-Tello BDC, Fonseca Aizpuru E, Alvarez-Troncoso J, Gonzalez A, Prieto-Gonzalez S, Freire M, Argibay AB, Pallares L, Todoli JA, Perez M, Bujan-Rivas S, Ibanez B; GEAS-SEMI Group. Efficacy and Safety of Anakinra Plus Standard of Care for Patients With Severe COVID-19: A Randomized Phase 2/3 Clinical Trial. JAMA Netw Open. 2023 Apr 3;6(4):e237243. doi: 10.1001/jamanetworkopen.2023.7243. PMID 37027155